CLINICAL TRIAL: NCT04061954
Title: Improving Family Cohesion Using a Comprehensive Family Program Addressing Parental Skills and Mental Health Issues in Traumatised Parents in Burundi
Brief Title: Umuryango Ukomera Uri Hamwe - Families Are Strong Together
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Konstanz (Other)
Collaborators: Vivo international e.V. (Industry); Psychologues sans Frontières Burundi (Other); Université Lumière de Bujumbura (Other)
Responsible Party: Principal Investigator, Anselm Crombach, Principal investigator, University of Konstanz
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UKCR19
Record Dates: First submitted 2019-08-17; First posted 2019-08-20 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Posttraumatic Stress Disorder; Aggressive Behaviour; Parental Maltreatment; Days Spent at the Landfill
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Aggression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Families in the intervention group received:
  1. Parents participate in a group intervention once a week for about 20 weeks, including psychoeducation on mental health and drug and alcohol abuse, anger management, family planning, parenting skills, communication skills, and dealing with couples conflicts
  2. Family visits to address topics as family cohesion, intra-familial communication and psychological basic need of children
  3. Trauma-focused therapies
  4. Parents receive training regarding agriculture and micro credit projects, and financial assistance
  5. One child per family receives a social skill training group preparing them for returning to school
  6. Access to schools and school material
  7. If needed medical assistance is provided
  8. If needed legal assistance is provided
  Interventions: Behavioral: Comprehensive family intervention including individual sessions of FORNET
- No intervention group (No Intervention): The control group was invited to participate in three interviews getting small amounts of money (~2,5 €) as decompensation of their time.

INTERVENTIONS:
Behavioral: Comprehensive family intervention including individual sessions of FORNET — Families in the intervention group received:
  1. Parents participate in a group intervention once a week for about 20 weeks, including psychoeducation on mental health and drug and alcohol abuse, anger management, family planning, parenting skills, communication skills, and dealing with couples conflicts
  2. Family visits to address topics as family cohesion, intra-familial communication and psychological basic need of children
  3. Trauma-focused therapies (FORNET), which aim also at reducing violent behaviour
  4. Parents receive training regarding agriculture and micro credit projects, and financial assistance
  5. One child per family receives a social skill training group preparing them for returning to school
  6. Access to schools and school material
  7. If needed medical assistance is provided
  8. If needed legal assistance is provided
  Arms: Intervention group

SUMMARY:
Children living in poverty often are at risk to leave their family to work at the landfill. The main reasons for this are torn family systems, family violence, exclusion, poverty and a lack of intra-familial communication. Children in the district of Buterere who spend their days on the streets or on the landfills of Bujumbura, Burundi to earn a living are particularly vulnerable. The project aims to create a safe environment for these young people and to strengthen their family structures in the long term. For this purpose, we plan to treat traumatized parents psychotherapeutically and to improve their parenting skills within the families in group and family sessions. The financial situation is to be improved in the medium term through agricultural group projects. In addition, participating children and youths will be granted access to school and education, and participate in a skill training group to improve social competencies. In the long term, parents are to set up savings and micro credit groups in order to ensure the education of the children. The project involves 40 families, which are particularly affected by poverty and traumatic experiences. The project is based on scientific findings of the implementing organizations, which carried out similar projects in Burundi in the last years.

DETAILED DESCRIPTION:
Children living in poverty often are at risk to leave their family to work at the landfill. The main reasons for this are torn family systems, family violence, exclusion, poverty and a lack of intra-familial communication. Psychological stress due to past political crises diminishes parents' ability to provide a safe environment for their children and often leads to maltreatment in the families. Children in the district of Buterere who spend their days on the streets or on the landfills of Bujumbura, Burundi to earn a living are particularly vulnerable. The project aims to create a safe environment for these young people and to strengthen their family structures in the long term to prevent them from losing family cohesion due to poverty and lack of support. For this purpose, we plan to treat traumatized parents psychotherapeutically and to improve their parenting skills within the families in group and family sessions. The individual trauma treatment aims also at reducing aggression problems frequently associated with trauma in order to reduce negative consequences for the children. The group sessions for parents aim to address subjects such as parenting skills, alcohol abuse, family planning, and conflicts amongst couples. The family visits aim at reinforcing communication between children and their parents. The financial situation is to be improved in the medium term through agricultural group projects. In addition, participating children and youths will be granted access to school and education, and participate in a skill training group. In the long term, parents are to set up savings and micro credit groups in order to ensure the education of the children. This multifactorial design should help to reduce the above-mentioned main risk factors for living on the street. The project involves 40 families, which are particularly affected by poverty and traumatic experiences. The legal guardians within the families are identified at the beginning of the project and directly involved to strengthen upbringing skills, to improve the economic situation of the family and to enable the adults affected by the violent political crises in Burundi to deal with their own psychological problems. In addition, one child between the ages of 5 and 20 per family is identified as the main beneficiary. This serves to gain a deeper insight into the family's communication and, in particular, to take sufficient account of the children's perspective. Through the integral approach of the project, which guarantees psychological, medical, social, legal and economic support, the children are to be protected from increasing violence on the streets and from family violence in the long term. The project is based on scientific findings of the implementing organizations, which carried out similar projects in Burundi in the last years.

ELIGIBILITY:
Inclusion Criteria:

* Parents who reported in a preliminary assessment to experience/or having experienced at least 3 of the following 5 conditions: (1) marital conflicts (2) difficulties to sleep in the past 4 weeks (3) Nightmares in the past 4 weeks (4) current social withdrawal (5) lost a loved one during the past year
* Parents who spend time at the landfill
* Parents with children between 7 and 16 who spend time at the landfill

Exclusion Criteria:

* Psychotic symptoms

Ages: 7 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-04-06 (Actual); Primary Completion 2020-05-27 (Actual); Study Completion 2020-05-27 (Actual)

PRIMARY OUTCOMES:
In parents: Change of load of traumatic symptoms measured via the PTSD Symptom Scale Interview for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) | baseline; 5 months follow-up; 9 months follow-up
  20 items assessing PTSD ranging from 0 - 4. Total sum score ranges from 0 to 80; sub scale intrusion: 0 - 20; sub scale avoidance: 0 - 8; sub scale negative cognitions: 0 - 28; sub scale hyperarousal: 0 - 24; higher values indicate more severe PTSD symptoms
In parents: Change of number of aggressive acts measured via an adaption of the Domestic and Community Violence | baseline; 5 months follow-up; 9 months follow-up
  32 items; answer categories: yes or no; sum score ranges from 0 - 32
In children: Change in experienced parental rejection measured via the short version of the Parental Acceptance Rejection Questionnaire | baseline; 5 months follow-up; 9 months follow-up
  24 items; answer categories: 1 - 4; sum score ranges from 24 - 96; the higher the more rejection
In children: Change of experienced parental maltreatment measured via a shortened version of the Maltreatment and Abuse Chronology of Exposure (MACE) | baseline; 5 months follow-up; 9 months follow-up
  total sum score ranges from 0 - 100; sum score of each sub scale ranges from 0 - 10
In children: Change of number of days spent at the landfill | baseline; 5 months follow-up; 9 months follow-up
  during the last 14 days; sum ranges from 0 - 14

CONTACTS AND LOCATIONS:
Locations (1):
- vivo international & Psychologues sans Frontières mental health center, Bujumbura, Bujumbura Mairie Province, Burundi

IPD SHARING:
Plan to Share IPD: No
Currently there is no plan to share individual participant data with other researchers not related to the institutions conducting the study. If data is shared, the PI will supervise those analyzing the data, e.g., students writing their theses.